CLINICAL TRIAL: NCT07285525
Title: Clinical Research Protocol on Accelerating Motor Rehabilitation in Postoperative Motor-Deficient Glioma Patients Using nrTMS
Brief Title: Accelerating Motor Recovery in Glioma Patients Using Postoperative nrTMS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRWEP2024W032040210; Beijing Municipal Health Commi (Other: Beijing Tiantan Hospital, Capital Medical University)
Record Dates: First submitted 2025-09-15; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Glioma
Keywords: Glioma; rehabilitation
MeSH Terms: conditions — Glioma | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham Comparator (Sham Comparator)
  Interventions: Device: sham stimulation
- nrTMS (Experimental)
  Interventions: Device: transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Device: transcranial magnetic stimulation (TMS) — Method for determining stimulation threshold: Using a positioning coil, based on the T1-3D MRI sequence and anatomical structure, single-pulse stimulation will be applied to the contralateral hand motor area. The stimulation intensity will be gradually increased from 50% until the action potential of the thenar eminence muscles exceeds 50 μV or until involuntary thumb movement occurs.
  High-frequency stimulation treatment:
  Localization of the ipsilateral thumb motor area: The positive points of intraoperative thumb motor area monitoring will be marked on the postoperative T1-3D image as the preferred target.
  Using the positioning coil, the target and surrounding areas will be stimulated, starting at 90% of the stimulation threshold intensity and increasing by 5% each time until involuntary thumb movement or an action potential of the thenar eminence muscles exceeding 50 μV is elicited. This point will be identified as the stimulation target.
  The treatment coil will be adjusted in angle
  Arms: nrTMS
Device: sham stimulation — Sham Stimulation Treatment:
  Target Localization: The same preferred target, based on the intraoperative thumb motor area monitoring points marked on the postoperative T1-3D image, will be used for coil placement to maintain consistency with the active treatment group.
  Stimulation Protocol: The sham treatment coil will be positioned over the ipsilateral thumb motor area. The stimulation will be delivered using parameters that replicate the auditory and somatosensory experience (e.g., clicking sound, scalp tapping) of real high-frequency nrTMS, but the magnetic field will be designed to not penetrate the cortex effectively. The intensity will be set to mimic the protocol of the active group (0% of a simulated threshold) without delivering neurologically effective stimulation. The coil angle may be adjusted to enhance the blinding by replicating the procedural steps of the active treatment.
  Arms: Sham Comparator

SUMMARY:
Project Name Clinical Research Protocol on Accelerating Motor Rehabilitation in Postoperative Motor-Deficient Glioma Patients Using nrTMS

Research Objectives

1. Investigate the relationship between motor rehabilitation and changes in motor functional networks after nrTMS therapy, and confirm the contralateral hand motor area as an effective rehabilitation target.
2. Validate the efficacy of high-frequency nrTMS stimulation in rehabilitating motor deficits in glioma patients.

Study Design > A randomized, double-blind, sham-controlled clinical trial. Eligible postoperative glioma patients with motor dysfunction will be randomized into nrTMS treatment or sham groups. High-frequency nrTMS or sham stimulation targeting the contralateral hand motor area will be administered for 7 consecutive days. Fugl-Meyer Assessment (FMA) scores and muscle strength of the affected limb will be evaluated to determine the superiority of nrTMS over sham stimulation.

Total Cases The study comprises two parts, each enrolling 43 patients.

Case Selection Inclusion Criteria:

A. Right-handed; B. Age: 25-65 years; C. No prior neurological disease history; D. Awake craniotomy with intraoperative direct cortical stimulation or MEP mapping for motor area localization; E. Postoperative pathology confirms newly diagnosed glioma; F. Willing to undergo nrTMS therapy; G. Persistent motor dysfunction (muscle strength/FMA score not restored to preoperative levels) at postoperative day 7.

Exclusion Criteria:

A. Tumor crossing midline to the contralateral hemisphere; B. Head motion >1 mm or rotation >1° during rs-fMRI acquisition; C. Absence of postoperative motor or speech dysfunction; D. Vulnerable populations (e.g., pregnant women). Treatment Protocol High-frequency nrTMS stimulation targeting the contralateral hand motor area (thumb region).

Efficacy Evaluation Primary Outcome: Muscle strength recovery rate of the affected limb.

Secondary Outcome: FMA score recovery rate. Safety Evaluation: Pre- and post-treatment MRI to monitor intracranial changes. Statistical Methods (1) Randomization into nrTMS and sham groups. (2) Baseline comparisons using t-tests and chi-square tests. (3) Longitudinal analysis of muscle strength (chi-square) and FMA scores (t-tests) at key timepoints: preoperative, pretreatment, post-treatment, 1/2/3 months postoperatively.

DETAILED DESCRIPTION:
Research Objectives:

Investigate the relationship between motor rehabilitation and changes in motor functional networks after nrTMS therapy, and confirm the contralateral hand motor area as an effective rehabilitation target.

Validate the efficacy of high-frequency nrTMS stimulation in rehabilitating motor deficits in glioma patients.

Study Design: A randomized, double-blind, sham-controlled clinical trial. Eligible postoperative glioma patients with motor dysfunction will be randomized into nrTMS treatment or sham groups. High-frequency nrTMS or sham stimulation targeting the contralateral hand motor area will be administered for 7 consecutive days. Fugl-Meyer Assessment (FMA) scores and muscle strength of the affected limb will be evaluated to determine the superiority of nrTMS over sham stimulation.

Total Cases: The study comprises two parts, each enrolling 43 patients.

Case Selection:

Inclusion Criteria:

A. Right-handed; B. Age: 25-65 years; C. No prior neurological disease history; D. Awake craniotomy with intraoperative direct cortical stimulation or MEP mapping for motor area localization; E. Postoperative pathology confirms newly diagnosed glioma; F. Willing to undergo nrTMS therapy; G. Persistent motor dysfunction (muscle strength/FMA score not restored to preoperative levels) at postoperative day 7.

Exclusion Criteria:

A. Tumor crossing midline to the contralateral hemisphere; B. Head motion >1 mm or rotation >1° during rs-fMRI acquisition; C. Absence of postoperative motor or speech dysfunction; D. Vulnerable populations (e.g., pregnant women).

Treatment Protocol: High-frequency nrTMS stimulation targeting the contralateral hand motor area (thumb region).

Efficacy Evaluation:

Primary Outcome: Muscle strength recovery rate of the affected limb. Secondary Outcome: FMA score recovery rate.

Safety Evaluation: Pre- and post-treatment MRI to monitor intracranial changes.

Statistical Methods:

1. Randomization into nrTMS and sham groups.
2. Baseline comparisons using t-tests and chi-square tests.
3. Longitudinal analysis of muscle strength (chi-square) and FMA scores (t-tests) at key timepoints: preoperative, pretreatment, post-treatment, 1/2/3 months postoperatively.

Detailed Description:

Project Title: Clinical Research Protocol: Accelerating Postoperative Motor Recovery in Patients with Motor Deficits after Glioma Surgery Using Navigated Repetitive Transcranial Magnetic Stimulation (nrTMS)

Research Objectives:

To reveal the relationship between motor recovery and changes in brain motor networks following nrTMS rehabilitation, and to confirm that the ipsilateral hand motor area is an effective target for motor rehabilitation.

To determine the effectiveness of high-frequency nrTMS stimulation in motor recovery for patients with motor deficits after glioma surgery.

Research Design: A randomized, double-blind, sham-controlled clinical trial will be conducted. Patients with motor deficits after glioma surgery who meet the inclusion/exclusion criteria will be randomly assigned to either the nrTMS treatment group or the sham stimulation group. The ipsilateral hand motor area will be targeted for high-frequency nrTMS or sham stimulation (7 working days). Motor recovery will be assessed using Fugl-Meyer Assessment (FMA) scores and muscle strength measurements to determine whether nrTMS is superior to sham stimulation in postoperative motor rehabilitation for glioma patients.

Total Number of Cases: The project will consist of two parts, with 43 patients in each part.

Case Selection:

Inclusion Criteria: A. Right-handed; B. Age: 25-65 years old; C. No history of neurological disease treatment before surgery; D. Patients underwent awake surgery with intraoperative direct cortical stimulation or intraoperative MEP and monopolar stimulation to identify the motor functional area; E. Postoperative pathology confirmed as newly diagnosed glioma; F. Eligible for nrTMS rehabilitation treatment; G. Motor function has not recovered to preoperative levels 7 days postoperatively, as indicated by muscle strength scores or FMA scores not returning to preoperative levels.

Exclusion Criteria: A. Tumor crossing the midline to the contralateral side; B. Head movement exceeding 1 mm or head rotation exceeding 1° during rs-fMRI data acquisition; C. Patients without postoperative motor or language motor deficits; D. Vulnerable or special populations, such as pregnant women.

Treatment Protocol: High-frequency nrTMS stimulation of the ipsilateral hand motor area (thumb motor area).

Efficacy Evaluation:

Primary Efficacy Indicators: Recovery rate of muscle strength in the affected limb.

Secondary Efficacy Indicators: Recovery rate of FMA scores.

Safety Evaluation Indicators: Pre- and post-treatment cranial MRI will be performed to confirm intracranial changes and ensure patient safety.

Statistical Methods:

All patients will be randomly divided into the nrTMS high-frequency stimulation group and the sham stimulation group.

Baseline data comparison: Depending on the data type, t-tests and chi-square tests will be used to compare baseline clinical data between the two groups, including gender, age, pathological type, pathological grade, and motor function status (muscle strength and FMA scores) at preoperative, pre-treatment, post-treatment, 1 month postoperative, 2 months postoperative, and 3 months postoperative.

Chi-square tests will be used to compare muscle strength recovery differences between the two groups at different time points.

Chi-square tests will also be used to compare muscle strength recovery differences within each group at different time points.

Independent-sample t-tests will be used to compare FMA score differences between the two groups at different time points.

Paired t-tests will be used to compare FMA score differences within each group at different time points.

Research Duration: October 2024 - October 2027

Research Background: Gliomas often invade motor areas of the brain, and their mass effect, along with damage to adjacent normal brain tissue during surgical resection, frequently leads to postoperative motor deficits in patients. Nearly 60% of patients with postoperative motor deficits fail to recover, resulting in permanent motor impairments that severely affect postoperative quality of life. Additionally, ample evidence indicates that gliomas, particularly low-grade gliomas, can induce cortical reorganization, enabling compensatory mechanisms for damaged functions. Therefore, stimulating motor function compensation and promoting cortical reorganization are critical for improving patient quality of life and prognosis.

Preliminary research by the investigators has shown that preoperative node efficiency in the hand motor area determines the recovery time for motor function in these patients. Gliomas growing in motor areas disrupt surrounding normal cortex, which participates in motor network reorganization to maintain normal motor function. However, surgical resection causes a "secondary" disruption to the already reorganized motor network. Node efficiency refers to a node's ability to transmit information within the motor network; higher node efficiency indicates a stronger role in the network. When the resection area is near the ipsilateral hand motor area, the node efficiency of the ipsilateral hand motor area has already increased due to cortical reorganization. Consequently, these patients inevitably experience postoperative motor deficits, with low recovery rates and prolonged recovery times.

Repetitive transcranial magnetic stimulation (rTMS) has been widely applied in the rehabilitation of neurological diseases and has been summarized in domestic and international clinical guidelines and expert consensus documents. However, in the clinical management and rehabilitation of glioma patients, TMS has only been used for preoperative mapping of motor and language functional areas, with no reports on its application for postoperative functional rehabilitation in glioma patients. This is because the rehabilitation targets and parameters used for stroke and other diseases are not entirely applicable to glioma patients, and there is a lack of clearly defined treatment targets between the two rehabilitation approaches.

Preliminary results from the research team suggest that high-frequency nrTMS stimulation of the ipsilateral hand motor area can significantly accelerate motor function recovery. However, due to the absence of a strict cohort-controlled trial, the reliability and effectiveness of nrTMS for motor recovery remain undetermined.

Domestic and International Research Status:

1.1 Glioma Growth Induces Cortical Reorganization and Alters Brain Functional Networks for Compensation Gliomas involving motor areas can cause severe motor deficits. However, patients often do not exhibit deficits preoperatively due to neuroplasticity and cortical reorganization. Unlike acute-onset strokes, gliomas are progressive, providing time for functional compensation. Traditional views suggest that compensation occurs concurrently with glioma development, first reorganizing peritumoral tissue and then recruiting distant ipsilateral and contralateral areas.

The hand motor area is crucial for motor regulation. The absence of preoperative deficits in some patients with gliomas in this area is due to glioma-induced cortical reorganization. Surgical resection causes "secondary" injury to the compensated cortex, leading to deficits. Subsequent recovery in some patients indicates that damaged function can be compensated again.

Gliomas can alter functional connectivity strength. Longitudinal studies show that functional recovery is accompanied by increased connectivity, linking brain functional reorganization to network changes. Graph theory analysis reveals topological property changes; for example, low-grade gliomas can increase shortest path length and decrease global efficiency in whole-brain networks. Preliminary work by the investigators indicates that glioma growth alters nearby functional networks, but the reorganization form varies, even for tumors in the same location, leading to diverse symptom presentations.

1.2 Damaged Functions Rely on Brain Functional Network Reorganization for Compensation Studies show that insular gliomas can compensate by increasing cortical thickness and gray matter volume of the contralateral insula. Analysis of whole-brain functional networks in insular glioma patients by the investigators indicated that left insular gliomas compensate by establishing new functional connections between the right insula and other left hemisphere regions, while right insular gliomas compensate by strengthening existing connections between the left insula and the right hemisphere.

Regarding motor networks, preliminary findings suggest that in early glioma growth, the tumor shortens the shortest path in the healthy motor network, sacrificing stability for compensation. As the glioma enlarges and damages the ipsilateral primary motor area more, the healthy network restores stability, maintaining motor function in the healthy hemisphere at lower transmission efficiency.

1.3 Postoperative Brain Functional Network Reorganization Is Key to Motor Recovery Research from Professor Duffau's team reported that during motor recovery, functional connectivity between the contralateral supplementary motor area (SMA) and the ipsilateral primary motor and sensory areas transitions from weak to strong, suggesting important roles for these areas. However, this study included only six patients with SMA gliomas and ignored hemispheric differences.

Preliminary experimental results from the investigators included 20 patients with postoperative motor deficits (10 nrTMS-sham, 10 nrTMS treatment). Comparison of node efficiency in the ipsilateral hand motor area at preoperative, 7 days postoperative, and recovery time points showed a significant decrease postoperatively and a significant increase upon recovery. The motor recovery rate was 90% in the nrTMS group versus 50% in the sham group. Thus, it is preliminarily concluded that high-frequency nrTMS stimulation of the ipsilateral hand motor area can effectively improve motor function, potentially by increasing node efficiency.

1.4 Principles and Applications of Repetitive Transcranial Magnetic Stimulation in Brain Function Recovery Transcranial magnetic stimulation (TMS) uses changing magnetic fields to generate electric fields for noninvasive cortical stimulation. Different frequency modes can produce excitatory (high-frequency, >1 Hz) or inhibitory (low-frequency, ≤1 Hz) effects. Long-term TMS can alter cortical excitability, reduce contralateral inhibition, enhance ipsilateral excitability, and promote cortical plasticity.

rTMS is widely used in clinical rehabilitation for post-stroke motor/language deficits, psychiatric disorders, and epilepsy, with guidelines and expert consensus available. However, in glioma patients, nrTMS has primarily been used for preoperative mapping, with few reports on postoperative functional rehabilitation. Some studies suggest nrTMS may aid recovery from acute ischemia after glioma surgery.

Therefore, this project aims to apply high-frequency nrTMS to the ipsilateral hand motor area using a double-blind, randomized, controlled design. Using rs-fMRI data and motor scores collected preoperatively, postoperatively (pre-nrTMS), and at recovery (post-nrTMS), the study will determine treatment effectiveness and investigate the mechanism: whether high-frequency stimulation accelerates the increase in node efficiency of the ipsilateral hand motor area, facilitating rapid motor recovery.

ELIGIBILITY:
Inclusion Criteria:

Right-handed.

Age between 25 and 65 years old.

No history of neurological disease treatment before surgery.

Underwent awake surgery with intraoperative direct cortical stimulation or motor evoked potential (MEP) mapping to identify the motor functional area.

Postoperative pathology confirmed as newly diagnosed glioma.

Eligible for navigated repetitive transcranial magnetic stimulation (nrTMS) rehabilitation treatment.

Persistent motor dysfunction (muscle strength or Fugl-Meyer Assessment (FMA) scores not returned to preoperative levels) at 7 days postoperatively.

Signed informed consent.

Exclusion Criteria:

Tumor crossing the midline to the contralateral hemisphere.

Excessive head motion (>1 mm translation or >1° rotation) during resting-state functional MRI (rs-fMRI) data acquisition.

Absence of postoperative motor or language motor deficits.

Vulnerable populations (e.g., pregnant women).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Muscle strength of the affected limb | muscle strength of the affected limb have returned to preoperative levels at pre-treatment, post-treatment, 1 month postoperative, 2 months postoperative, and 3 months postoperative.
  Motor function recovery is defined as the affected limb's muscle strength returning to preoperative levels.

SECONDARY OUTCOMES:
Rate of Fugl-Meyer Assessment (FMA) Score Recovery for the Affected Upper Limb | Assessed at pre-treatment (postoperative day 7), post-treatment (after 7 days of intervention), 1 month, 2 months, and 3 months postoperatively.
  Recovery is defined as the FMA score for the affected upper limb returning to the preoperative level.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, None Selected, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Potgieser AR, de Jong BM, Wagemakers M, Hoving EW, Groen RJ. Insights from the supplementary motor area syndrome in balancing movement initiation and inhibition. Front Hum Neurosci 2014;8:960. 2. Morone G, Capone F, Iosa M, et al. May Dual Transcranial Direct Current Stimulation Enhance the Efficacy of Robot-Assisted Therapy for Promoting Upper Limb Recovery in Chronic Stroke? Neurorehabil Neural Repair 2022;36:800-809. 3. Youssef H, Mohamed NAE, Hamdy M. Comparison of bihemispheric and unihemispheric M1 transcranial direct current stimulations during physical therapy in subacute stroke patients: A randomized controlled trial. Neurophysiol Clin 2023;53:102895. 4. Bikson M, Hanlon CA, Woods AJ, et al. Guidelines for TMS/tES clinical services and research through the COVID-19 pandemic. Brain Stimul 2020;13:1124-1149. 5. Steeves T, McKinlay BD, Gorman D, et al. Canadian guidelines for the evidence-based treatment of tic disorders: behavioural therapy, deep brain stimulation, and transcranial magnetic stimulation. Can J Psychiatry 2012;57:144-151. 6. 中国医师协会神经调控专业委员会电休克与神经刺激学组. 重复经颅磁刺激治疗专家共识. 转化医学杂志 2018;7:4-9. 7. Krieg SM, Shiban E, Buchmann N, et al. Utility of presurgical navigated transcranial magnetic brain stimulation for the resection of tumors in eloquent motor areas. J Neurosurg 2012;116:994-1001. 8. 王引言, 方晟宇, 李连旺, et al. 重复经颅磁刺激治疗脑胶质瘤术后运动功能障碍的临床分析(附五例报告). 中华神经外科杂志 2020;36:458-462. 9. Herbet G, Maheu M, Costi E, Lafargue G, Duffau H. Mapping neuroplastic potential in brain-damaged patients. Brain : a journal of neurology 2016;139:829-844. 10. Almairac F, Duffau H, Herbet G. Contralesional macrostructural plasticity of the insular cortex in glioma patients. Neurology 2018:1. 11. Duffau H. Functional Mapping before and after Low-Grade Glioma Surgery: A New Way to Decipher Various Spatiotemporal Patterns of Individual Neuroplastic Potential in Brain Tumor Patients. Cancers (Basel) 2020;12. 12. Duffau H. Hodotopy, neuroplasticity and diffuse gliomas. Neurochirurg